CLINICAL TRIAL: NCT04090268
Title: Precision Exercise Program in Children With Malignant Hemopathies Undergoing Therapy and/or Hematopoietic Stem Cell Transplantation: The "Sport Therapy" Project
Brief Title: Precision Exercise in Children With Malignant Hemopathies
Acronym: SportTherapy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Milano Bicocca (Other)
Collaborators: Comitato Maria Letizia Verga,Italy (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 284 BIONDI
Record Dates: First submitted 2019-06-02; First posted 2019-09-16 (Actual); Last update posted 2024-01-02 (Actual); Status verified 2023-12

CONDITIONS: Leukemia, Myeloid, Acute; Leukemia, B-cell; Leukemia, T Cell; Lymphoma, Hodgkin; Lymphoma, Non-Hodgkin; Drepanocytosis; Thalassemia Major; Adrenoleukodystrophy
Keywords: exercise; children; adolescent; cancer; malignant hemopathies; leukemia; lymphoma; hematopoietic stem cell transplant; survivor; oxidative metabolism; strength; balance; flexibility; quality of life
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Leukemia, B-Cell; Leukemia, T-Cell; Hodgkin Disease; Lymphoma, Non-Hodgkin; Sickle Cell Trait; beta-Thalassemia; Adrenoleukodystrophy; Motor Activity; Neoplasms; Leukemia; Lymphoma

STUDY DESIGN:
Intervention Model Description: Analytical study, stratified, evaluating the impact of a non-pharmacological treatment (training)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Children with malignant hemopathies (Experimental): Children with malignant hemopathies attending a precision exercise training
  Interventions: Other: Sport Therapy
- Healthy children (No Intervention): Healthy children

INTERVENTIONS:
Other: Sport Therapy — Children and adolescent with malignant hemopathies will attend a 3 days/weekly combined training
  Other Names: Precision exercise program
  Arms: Children with malignant hemopathies

SUMMARY:
In the early years of life and during adolescence, physical activity is crucial for good development of motor skills. It is even more so for those children and young people who are forced to undergo anti-cancer therapies and therefore undergo long periods of hospitalization (often bedridden) and prolonged periods of physical inactivity.

The research project "Sport Therapy" was born with the aim of demonstrating that, through targeted physical activity administered by the sports physician in collaboration with the pediatrician hematologist, it is possible to facilitate the full recovery of these patients, avoiding the high risk of chronic diseases related to a sedentary lifestyle and allowing them to better reintegrate, once healed, in their community of origin (school, sport and social relations).

The research project "Sport Therapy" was born within the Maria Letizia Verga Center at the Pediatric Clinic of the University of Milan Bicocca, at the Foundation for the Mother and Her Child, San Gerardo Hospital in Monza. Every year, around 80 children and adolescents with leukemia, lymphoma or blood disorders leading to bone marrow transplantation are treated here.

DETAILED DESCRIPTION:
State of the art. Today, thanks to the progress made in the early diagnosis and treatment of cancer, there are more than 300 thousand young patients in Europe who have been cured of pediatric cancer, and by 2020 there will be almost half a million . For these children and young people, having the opportunity to perform targeted physical activity during treatment plays a key role in preventing diseases due to physical inactivity, which are one of the worst and most widespread consequences for healed patients.

Children and adolescents suffering from cancer of the blood, because of the therapies to which they are subjected, suffer a progressive reduction in respiratory and cardiac capacity, as well as muscle strength. Targeted physical exercise is a possible therapeutic approach to solving their significant problems of reduced ability to perform exercise. It is possible to administer this type of therapy thanks to the synergy created by the collaboration between pediatricians, hematologists, and sports physicians.

Why is this research important? For at least three reasons:

1. the results of the "Sport Therapy" research project will launch precision training as one of the therapeutic weapons available to combat the consequences of hematological diseases in childhood;
2. by increasing the physical capacity of children and adolescents with malignant hemopathies during the phases of cancer treatment, the investigators will reduce the heavy legacy left by treatment, thus bridging the gap regarding their disadvantage towards healthy peers and ensuring their full reintegration into their communities (school, sport, social relations);
3. a standardization of the methodology for using precision exercise in hospitalized children and adolescents will facilitate the monitoring of the progress of these type of interventions at the international level and the data from the "Sport Therapy" project will allow governments and concerned bodies not to further postpone the establishment of strategies necessary to improve the health and welfare of people cured of cancer diseases.

Innovative aspects of research. At the end of the research project "Sport Therapy":

* new strategies will be available to combat cardiopulmonary and skeletal muscle damage resulting from anticancer therapies;
* it will be definitively demonstrated how, from the very beginning of the disease, physical exercise can be a therapeutic option and not just a decorative element in the critical process of caring for children and adolescents suffering from oncological blood diseases, from the beginning of the disease;
* the possibility of introducing new technical figures in the hospital context will be clear. Sports medicine physician and exercise physiologists will be part of the multidisciplinary team that connects the hospital environment to the territory;
* the future perspective, once the experimentation has been completed and the effectiveness of the precision training intervention on the psycho-physical health of children and adolescents suffering from cancer has been demonstrated, will be to make "Sport Therapy" a permanent care service during the treatment of patients of developing age.

ELIGIBILITY:
Inclusion Criteria:

* Children with malignant hemopathies attending the Maria Letizia Verga Center

Exclusion Criteria:

* Children under 2 years

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 380 (Estimated)
Dates: Start 2017-04-03 (Actual); Primary Completion 2025-04-03 (Estimated); Study Completion 2026-04-03 (Estimated)

PRIMARY OUTCOMES:
Change from baseline oxidative metabolism at 12 weeks | 12 weeks
  Maximal O2 uptake and skeletal muscle O2 extraction
Change from baseline strength of upper and lower limbs (1RM) at 12 weeks | 12 weeks
  1 repetition maximal
Change from baseline balance at 12 weeks | 12 weeks
  Stabilometry
Change from baseline Quality of Life questionnaire at 12 weeks | 12 weeks
  The PedsQL Measurement Model is a modular approach to measuring health-related quality of life in healthy children and adolescents and those with acute and chronic health conditions. The PedsQL Measurement Model integrates seamlessly both generic core scales and disease-specific modules into one measurement system. The 23-item PedsQL Generic Core Scales were designed to measure the core dimensions of health as delineated by the World Health Organization, as well as role (school) functioning. The 4 Multidimensional Scales (physical, emotional, social, school) and 3 Summary Scores (physical health, psycho-social health and total). Each item has a score between 0 and 4, so the scale score is between 0-100. Higher scores indicate a better QoL.

SECONDARY OUTCOMES:
Change from baseline Satisfaction at 12 weeks | 12 weeks
  Visual analog scale (VAS), from 0 to 10, where 0 is any satisfaction and 10 maximal satisfaction.
Change from baseline 6 minute walking test at 12 weeks | 12 weeks
  6 minute walking test
Change from baseline Time up and down stairs test at 12 weeks | 12 weeks
  Time up and down stairs test
Change from baseline yo yo test at 12 weeks | 12 weeks
  Shuttle incremental walking/run test
Change from baseline MOON test at 12 weeks | 12 weeks
  MOON test

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Biondi, MD, PhD, Principal Investigator — University of Milano Bicocca
Locations (1):
- Maria Letizia Verga Center, Pediatric Clinic, University of Milan Bicocca, at the Foundation for the Mother and Her Child, Monza, MB, Italy

IPD SHARING:
Plan to Share IPD: Yes
Oxidative metabolism and MOON test variables will be shared with other colleagues involved in similar research protocols
Supporting Information: SAP, ICF
Time Frame: In July 2019 data will be shared, forever
Access Criteria: Invitation of a common folder in google drive
URL: https://drive.google.com/drive/u/0/folders

REFERENCES:
- [Background] Lanfranconi F, Pollastri L, Ferri A, Fraschini D, Masera G, Miserocchi G. Near infrared spectroscopy (NIRS) as a new non-invasive tool to detect oxidative skeletal muscle impairment in children survived to acute lymphoblastic leukaemia. PLoS One. 2014 Jun 23;9(6):e99282. doi: 10.1371/journal.pone.0099282. eCollection 2014. PMID 24956391
- [Background] Arico M, Valsecchi MG, Rizzari C, Barisone E, Biondi A, Casale F, Locatelli F, Lo Nigro L, Luciani M, Messina C, Micalizzi C, Parasole R, Pession A, Santoro N, Testi AM, Silvestri D, Basso G, Masera G, Conter V. Long-term results of the AIEOP-ALL-95 Trial for Childhood Acute Lymphoblastic Leukemia: insight on the prognostic value of DNA index in the framework of Berlin-Frankfurt-Muenster based chemotherapy. J Clin Oncol. 2008 Jan 10;26(2):283-9. doi: 10.1200/JCO.2007.12.3927. PMID 18182669
- [Background] Aznar S, Webster AL, San Juan AF, Chamorro-Vina C, Mate-Munoz JL, Moral S, Perez M, Garcia-Castro J, Ramirez M, Madero L, Lucia A. Physical activity during treatment in children with leukemia: a pilot study. Appl Physiol Nutr Metab. 2006 Aug;31(4):407-13. doi: 10.1139/h06-014. PMID 16900230
- [Background] Bangsbo J, Iaia FM, Krustrup P. The Yo-Yo intermittent recovery test : a useful tool for evaluation of physical performance in intermittent sports. Sports Med. 2008;38(1):37-51. doi: 10.2165/00007256-200838010-00004. PMID 18081366
- [Background] Geiger R, Strasak A, Treml B, Gasser K, Kleinsasser A, Fischer V, Geiger H, Loeckinger A, Stein JI. Six-minute walk test in children and adolescents. J Pediatr. 2007 Apr;150(4):395-9, 399.e1-2. doi: 10.1016/j.jpeds.2006.12.052. PMID 17382117
- [Background] Gohar SF, Comito M, Price J, Marchese V. Feasibility and parent satisfaction of a physical therapy intervention program for children with acute lymphoblastic leukemia in the first 6 months of medical treatment. Pediatr Blood Cancer. 2011 May;56(5):799-804. doi: 10.1002/pbc.22713. Epub 2011 Jan 16. PMID 21370414
- [Background] Gotte M, Kesting S, Albrecht C, Worth A, Bos K, Boos J. MOON-test - determination of motor performance in the pediatric oncology. Klin Padiatr. 2013 May;225(3):133-7. doi: 10.1055/s-0033-1343411. Epub 2013 Apr 18. PMID 23599231
- [Background] Hartman A, te Winkel ML, van Beek RD, de Muinck Keizer-Schrama SM, Kemper HC, Hop WC, van den Heuvel-Eibrink MM, Pieters R. A randomized trial investigating an exercise program to prevent reduction of bone mineral density and impairment of motor performance during treatment for childhood acute lymphoblastic leukemia. Pediatr Blood Cancer. 2009 Jul;53(1):64-71. doi: 10.1002/pbc.21942. PMID 19283791
- [Background] Haupt R, Spinetta JJ, Ban I, Barr RD, Beck JD, Byrne J, Calaminus G, Coenen E, Chesler M, D'Angio GJ, Eiser C, Feldges A, Gibson F, Lackner H, Masera G, Massimo L, Magyarosy E, Otten J, Reaman G, Valsecchi MG, Veerman AJ, Penn A, Thorvildsen A, van den Bos C, Jankovic M; International Berlin-Frankfurt-Munster Study Group Early and Late Toxicity Educational Committee (I-BFM-SG ELTEC). Long term survivors of childhood cancer: cure and care. The Erice statement. Eur J Cancer. 2007 Aug;43(12):1778-80. doi: 10.1016/j.ejca.2007.04.015. Epub 2007 May 31. PMID 17543517
- [Background] Hogarty AN, Leahey A, Zhao H, Hogarty MD, Bunin N, Cnaan A, Paridon SM. Longitudinal evaluation of cardiopulmonary performance during exercise after bone marrow transplantation in children. J Pediatr. 2000 Mar;136(3):311-7. doi: 10.1067/mpd.2000.103444. PMID 10700686
- [Background] Jenney ME, Faragher EB, Jones PH, Woodcock A. Lung function and exercise capacity in survivors of childhood leukaemia. Med Pediatr Oncol. 1995 Apr;24(4):222-30. doi: 10.1002/mpo.2950240403. PMID 7700166
- [Background] San Juan AF, Fleck SJ, Chamorro-Vina C, Mate-Munoz JL, Moral S, Perez M, Cardona C, Del Valle MF, Hernandez M, Ramirez M, Madero L, Lucia A. Effects of an intrahospital exercise program intervention for children with leukemia. Med Sci Sports Exerc. 2007 Jan;39(1):13-21. doi: 10.1249/01.mss.0000240326.54147.fc. PMID 17218878
- [Background] San Juan AF, Fleck SJ, Chamorro-Vina C, Mate-Munoz JL, Moral S, Garcia-Castro J, Ramirez M, Madero L, Lucia A. Early-phase adaptations to intrahospital training in strength and functional mobility of children with leukemia. J Strength Cond Res. 2007 Feb;21(1):173-7. doi: 10.1519/00124278-200702000-00031. PMID 17313277
- [Background] Lucia A, Ramirez M, San Juan AF, Fleck SJ, Garcia-Castro J, Madero L. Intrahospital supervised exercise training: a complementary tool in the therapeutic armamentarium against childhood leukemia. Leukemia. 2005 Aug;19(8):1334-7. doi: 10.1038/sj.leu.2403799. No abstract available. PMID 15931268
- [Background] Maggiani A, Tremolizzo L, Della Valentina A, Mapelli L, Sosio S, Milano V, Bianchi M, Badi F, Lavazza C, Grandini M, Corna G, Prometti P, Lunetta C, Riva N, Ferri A, Lanfranconi F; ME&SLA Study #. Osteopathic Manual Treatment for Amyotrophic Lateral Sclerosis: A Feasibility Pilot Study. Open Neurol J. 2016 Aug 26;10:59-66. doi: 10.2174/1874205X01610010059. eCollection 2016. PMID 27651843
- [Background] Nagashima T, Sato F, Chuma T, Mano Y, Sasaki I, Mori M, Higa T, Masauji N, Kasai M, Orba Y, Shinohara T, Nagashima K. Chronic demyelinating polyneuropathy in graft-versus-host disease following allogeneic bone marrow transplantation. Neuropathology. 2002 Mar;22(1):1-8. PMID 12030409
- [Background] Tan SY, Poh BK, Chong HX, Ismail MN, Rahman J, Zarina AL, Juraida AR, Tahir A, Ruzita AT, Roslee R, Shanita SN, Hamidah A, Shah MI, Norimah AK. Physical activity of pediatric patients with acute leukemia undergoing induction or consolidation chemotherapy. Leuk Res. 2013 Jan;37(1):14-20. doi: 10.1016/j.leukres.2012.09.005. Epub 2012 Oct 23. PMID 23099236
- [Background] Zaino CA, Marchese VG, Westcott SL. Timed up and down stairs test: preliminary reliability and validity of a new measure of functional mobility. Pediatr Phys Ther. 2004 Summer;16(2):90-8. doi: 10.1097/01.PEP.0000127564.08922.6A. PMID 17057533
- See also: Sport Therapy project page — https://comitatomarialetiziaverga.it/care-and-therapy/sport-therapy/